CLINICAL TRIAL: NCT06318442
Title: How GLP-1 Analogues Prevent Steroid-Induced Diabetes
Brief Title: The GAPSID Study - How GLP-1 Analogues Prevent Steroid-Induced Diabetes
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Imperial College London (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Basic Science
Other Study IDs: 22HH8018
Record Dates: First submitted 2024-03-06; First posted 2024-03-19 (Actual); Last update posted 2024-10-02 (Actual); Status verified 2024-09

CONDITIONS: Steroid-Induced Diabetes; Steroid Induced Hyperglycemia
MeSH Terms: interventions — Metformin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Once daily semaglutide (Experimental): Once daily semaglutide 3 mg (uptitrated to 3 mg twice daily after two days).
  Interventions: Drug: Semaglutide Oral Product
- - Metformin (Active Comparator): Metformin modified release tablets (500mg once daily for the first two days, then 500 mg twice daily).
  Interventions: Drug: Metformin Oral Tablet
- Placebo (Placebo Comparator): Placebo tablets
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Semaglutide Oral Product — Oral semaglutide 3mg once uptitrated to twice daily
  Arms: Once daily semaglutide
Drug: Metformin Oral Tablet — Metformin modified release tablets 500mg once daily uptitrated to twice daily).
  Arms: - Metformin
Drug: Placebo — Placebo tablets
  Arms: Placebo

SUMMARY:
TITLE: How GLP-1 Analogues prevent steroid-induced diabetes (The GAPSID Study)

DESIGN: A double-blind study evaluating how GLP-1 analogues, compared with metformin, prevent hyperglycaemia in response to a 7-day course of dexamethasone (DEX) 6 mg once daily. This is a mechanistic experimental medicine study.

AIMS: To evaluate the mechanisms by which GLP-1 analogues reduce steroid-induced hyperglycaemia compared to metformin.

OUTCOME MEASURES:

* Primary: Glucose tolerance in response to standardised mixed meal test (MMT) lasting for 240 minutes, measured in all participants at baseline and on day 7 DEX.
* Secondary: Indices of insulin resistance (M-value), beta-cell function (acute insulin response to glucose) and disposition, as measured by a combined IV glucose tolerance test and hyperinsulinaemic-euglycaemic clamp, performed at baseline and on day 7 DEX.
* Exploratory: Tissue specific changes in adipose AMPK determined from adipose and muscle biopsies, taken from a subset of approximately 8 individuals in each group.

ELIGIBILITY: People living with pre-diabetes or lifestyle controlled diabetes

STUDY DURATION: This study will take place over 3 weeks for each partcipant. Study procedures include 10 days of baseline continuous glucose monitoring (CGM) followed by 7 days of dexamethasone with GLP-1, metformin or placebo. Participants will attend a follow-up visit 3-5 days after completing the 7-day course of study drug. The study will run over a period of 3 years.

ANTICIPATED IMPACT: Mechanistic evidence for the use of GLP-1 analogues, compared with metformin, in the treatment of steroid-induced diabetes.

ELIGIBILITY:
Inclusion Criteria:

* Adults ≥ 18 years;
* Male or female;
* Pre-diabetes (HbA1c ≥42 and <47 mmol/mol, or lifestyle-controlled diabetes (HbA1c ≥48 and ≤52 mmol/mol); measurements within range on two separate occasions ≥90 days apart)
* Body mass index ≥22.5 kg/m2

Exclusion Criteria:

* Prior treatment with any diabetes medication within 90 days;
* Current or planned pregnancy, or current breastfeeding;
* Previous treatment with GC (topical, oral, injected) within 30 days or 90 days for extended-release injected GCs (e.g. Depo-Medrone);
* Continuing requirement for GC treatment (e.g. for steroid replacement, chronic inflammatory or immunological condition);
* Treatment with medications altering DEX pharmacokinetics (e.g. phenytoin, carbamazepine, ritonavir).
* History of pancreatitis, renal disease (eGFR <30), severe hepatic impairment, gallbladder disorders, or GI disease (e.g. IBD), heart failure, history of medullary thyroid cancer (MTC), or previous skin reactions.
* History of bleeding disorders of anticoagulant therapies (exclusion from the biopsy substudy only)
* History of giving blood or having taken part in another non-related study in the last three months
* History of any other medical, psychological condition, or use of any medications, which, in the opinion of the investigators, would either interfere with the study or compromise the safety of the participant.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2024-05-15 (Actual); Primary Completion 2027-06-01 (Estimated); Study Completion 2027-06-01 (Estimated)

PRIMARY OUTCOMES:
Difference in Glucose tolerance | Through study completion, on day 7 dexamethasone and study medication
  Glucose tolerance as measured by glucose area under the curve (AUC), in response to standardised mixed meal test (MMT) lasting for 240 minutes. This will be measured in all participants at baseline and at the end of the study medication period (after 7 days of dexamethasone and study medication).

SECONDARY OUTCOMES:
Difference in insulin secretion | Day 6 of dexamethasone and study medication
  This will be measured by the acute insulin response to glucose based on the incremental AUC for insulin during the first 10 minutes of an IVGTT and the second phase insulin response based on incremental AUC for insulin during +10 to +60 minutes.
  This will be measured in a subset of patients (10 from each randomisation group), performed at baseline and on day 6 of dexamethasone and study medication
Difference in insulin sensitivity | Day 6
  This will be measured by the M value, based on the glucose infusion rate during the last 60 minutes of a hyperinsulinaemic-euglycaemic clamp.
  This will be measured in a subset of patients (10 from each randomisation group), performed at baseline and on day 6 of dexamethasone and study medication
Difference in insulin sensitivity | Day 6
  This will be measured by the M/I index, calculated by the M value divided by the mean steady state insulin levels during the last 60 minutes of a hyperinsulinaemic-euglycaemic clamp.
  This will be measured in a subset of patients (10 from each randomisation group), performed at baseline and on day 6 of dexamethasone and study medication
Difference in insulin sensitivity | Day 6
  This will be measured by the disposition index. This will be calculated as the product of the AIRg and M value during the combined IVGTT and hyperinsulinaemic-euglycaemic clamp.
  This will be measured in a subset of patients (10 from each randomisation group), performed at baseline and on day 6 of dexamethasone and study medication.

OTHER OUTCOMES:
Mean glucose and glycaemic variation by continuous glucose monitoring (CGM), using a validated blinded system (Dexcom G7). | Through study completion
  A baseline recording will be made for 10 days prior to DEX. A second 10-day recording will be made covering the 7 days of DEX and for 3 days after.
Changes in fasting gut hormones | Through study completion, on day 7 dexamethasone and study medication
  Fasting glucose will be measured at baseline and after a 7-day course of DEX and treatment intervention.
Changes in fasting gut hormones | Through study completion, on day 7 dexamethasone and study medication
  Fasting insulin and c-peptide levels will be measured at baseline and after a 7-day course of DEX and treatment intervention.
Changes in fasting gut hormones | Through study completion, on day 7 dexamethasone and study medication
  Fasting glucagon levels will be measured at baseline and after a 7-day course of DEX and treatment intervention.
Changes in fasting lipid profile | Through study completion, on day 7 dexamethasone and study medication
  Fasting lipid profiles will be measured at baseline and after a 7-day course of DEX and treatment intervention.
Changes in post prandial gut hormones | Through study completion, on day 7 dexamethasone and study medication
  Post prandial insulin and c-peptide levels will be measured during the mixed meal test, performed at baseline and after a 7-day course of DEX and treatment intervention.
Changes in post prandial gut hormones | Through study completion, on day 7 dexamethasone and study medication
  Post prandial glucagon levels will be measured during the mixed meal test, performed at baseline and after a 7-day course of DEX and treatment intervention.
Changes in anthropometrics | Through study completion, on day 7 dexamethasone and study medication
  Anthropometric measurements of height and weight will be combined to report BMI kg/m2 before and after a 7-day course of DEX and treatment intervention.
Changes in anthropometrics | Through study completion, on day 7 dexamethasone and study medication
  Measurements of hip and waist circumference will be combined to calculate the waist:hip ratio before and after a 7-day course of DEX and treatment intervention.
Tissue specific changes in AMPK determined from adipose and muscle biopsies | Through study completion, on day 7 dexamethasone and study medication
  This will be taken from a subset of approximately 8 individuals in each group prior to, and at the end of a 7 day course of DEX. Depending on emerging data and participant uptake, this may be subject to change.

CONTACTS AND LOCATIONS:
Overall Officials: Karim Meeran, Principal Investigator — Imperial College London
Locations (1):
- Imperial College Healthcare NHS Trust, London, United Kingdom